CLINICAL TRIAL: NCT06943534
Title: Omalizumab Weight-Based Dosing Efficacy Trial
Acronym: OWED-T
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Wayne G. Shreffler, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025P000538
Record Dates: First submitted 2025-03-28; First posted 2025-04-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Allergies; Food Allergy
Keywords: omalizumab
MeSH Terms: conditions — Hypersensitivity; Food Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients Receiving 5mg/kg of omalizumab (Active Comparator): Participants randomized to this arm will receive a does of 5mg/kg Omalizumab per month divided every two (2) weeks for 16 weeks.
  Interventions: Drug: 5mg/kg omalizumab injection
- Patients Receiving 15mg/kg of omalizumab (Active Comparator): Participants randomized to this arm will receive a does of 15mg/kg Omalizumab per month divided every two (2) weeks for 16 weeks.
  Interventions: Drug: 15mg/kg omalizumab injection

INTERVENTIONS:
Drug: 5mg/kg omalizumab injection — 5mg/kg of omalizumab
  Other Names: Xolair
  Arms: Patients Receiving 5mg/kg of omalizumab
Drug: 15mg/kg omalizumab injection — 15mg/kg of omalizumab
  Other Names: Xolair
  Arms: Patients Receiving 15mg/kg of omalizumab

SUMMARY:
This research is being conducted to assess the safety and effectiveness of increased dosing of Omalizumab for food allergies.

DETAILED DESCRIPTION:
This research is being conducted to assess the safety and effectiveness of omalizumab for food allergies dosed differently from what is currently FDA approved. The study hypothesizes the current way of dosing omalizumab may not work well for all patients with food allergy and it unnecessarily excludes some individuals with very high allergic antibody (IgE) who may benefit. This study will include subjects regardless of IgE level. One of the goals is to learn more about how safe and effective Omalizumab is for people with these high IgE levels, since this has not been fully studied before.

ELIGIBILITY:
Inclusion Criteria:

* A positive prick skin test (PST) with a wheal ≥ 6 mm to at least two of the relevant foods (peanut, cashew, walnut, egg, or milk)
* Positive food specific IgE (≥2.0 kUA/L) to at least two of the relevant foods
* A positive history of clinical reaction to at least one of the qualifying foods other than the challenge-qualifying food

(If meeting above criteria):

* Positive oral food challenge (OFC) to one of the potentially qualifying foods at a cumulative dose of ≤144 mg (maximum tolerated dose ≤30 mg)

Exclusion Criteria:

* Weight >80 kg at time of screening
* Clinically significant laboratory abnormalities at screening.
* Sensitivity or suspected/known allergy to any ingredients (including excipients) of omalizumab.
* Poorly controlled or severe asthma/wheezing at screening
* History of severe anaphylaxis to participant-specific foods that will be used in this study, defined as neurological compromise, PICU admission f for continuous epinephrine for hypotension or severe respiratory compromise requiring intubation.
* Treatment with a burst of oral, intramuscular (IM), or intravenous (IV) steroids of more than two days for an indication other than asthma/wheezing within 30 days of screening.
* Currently receiving oral, IM, or IV corticosteroids, tricyclic antidepressants, or β-blockers.
* Past or current history of eosinophilic gastrointestinal disease within three years of screening.
* Past or current history of cancer, or currently being investigated for possible cancer.
* Past or current history of any food immunotherapy (e.g., OIT, SLIT, EPIT) within 6 months of screening.
* Treatment with monoclonal antibody therapy, or other immunomodulatory therapy within 6 months of screening.
* Inability to discontinue antihistamines for minimum wash-out periods required for SPTs or OFCs.
* Pregnant or breastfeeding or intending to become pregnant during the study.
* Evidence of clinically significant chronic disease.

Ages: 1 Year to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants that tolerate the 600 mg dose after treatment. | 16 Weeks
  The primary analysis of outcome is on the proportion of subjects tolerating at least 600 mg at the post-treatment OFC in either group against the expected outcome without treatment based on OUTMATCH data.

SECONDARY OUTCOMES:
Other measures of omalizumab treatment effect on food allergy | 16 Weeks
  Secondary efficacy endpoint analysis will also be determined at OFC following 16-weeks of treatment:
  ● The proportion of participants that tolerate a single dose 1000 mg allergen
Other measures of omalizumab treatment effect on food allergy | 16 Weeks
  Secondary efficacy endpoint analysis will also be determined at OFC following 16-weeks of treatment:
  ● The proportion of participants that tolerate a single dose 2000 mg allergen
Other measures of omalizumab treatment effect on food allergy | 16 Weeks
  Secondary efficacy endpoint analysis will also be determined at OFC following 16-weeks of treatment:
  ● The proportion of participants that tolerate two doses of 2000 mg allergen
Other measures of omalizumab treatment effect on food allergy | 16 Weeks
  Secondary efficacy endpoint analysis will also be determined at OFC following 16-weeks of treatment:
  ● Reaction severity of positive post treatment reactions using the CoFAR grading scale ranging from 1 (mild) to 5 (death)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Shreffler, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No